CLINICAL TRIAL: NCT00203229
Title: A Double-Blind Placebo Controlled Add-on Study to Determine the Efficacy and Safety of Lamictal (Lamotrigine) in Patients With Trigeminal Neuralgia (Tic Doloureux)
Brief Title: Research Study to Test Safety and Effectiveness of Investigational Drug in Patients With Trigeminal Neuralgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MAS/LAM101; H92001 (Other Grant/Funding Number: GlaxoSmithKline)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-05

CONDITIONS: Trigeminal Neuralgia
Keywords: Double-Blind; Placebo-Controlled
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — Lamotrigine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Dosing Schedule Morning Evening Daily Total Week 1-2 ---- 50mg 50mg Week 3-4 50mg 50mg 100mg Week 5 100mg 100mg 200mg Week 6 150mg 150mg 300mg Week 7 200mg 200mg 400mg Week 8 (if needed for pain) 200mg 300mg 500mg Week 9 (if needed for pain) 300mg 300mg 600mg Week 10 (if needed for pain) 300mg 400mg 700mg
  Interventions: Drug: Placebo
- Lamotrigine (Active Comparator): Dosing Schedule Morning Evening Daily Total Week 1-2 ---- 50mg 50mg Week 3-4 50mg 50mg 100mg Week 5 100mg 100mg 200mg Week 6 150mg 150mg 300mg Week 7 200mg 200mg 400mg Week 8 (if needed for pain) 200mg 300mg 500mg Week 9 (if needed for pain) 300mg 300mg 600mg Week 10 (if needed for pain) 300mg 400mg 700mg
  Interventions: Drug: lamotrigine

INTERVENTIONS:
Drug: lamotrigine — The intervention type is 'drug' and this arm is a placebo pill created and supplied by the manufacturers of lamotrigine (Lamictal). This drug is an anti-seizure medication.
  Other Names: Lamictal; Lamictal XR
  Arms: Lamotrigine
Drug: Placebo — The intervention type is 'drug' and this arm is a placebo pill created and supplied by the manufacturers of lamotrigine (Lamictal) to be exact replicas of the actual drug being studied. The placebo arm is titrated in the exact same manor as the active drug arm.
  Arms: Placebo

SUMMARY:
This research study will look at the safety (e.g., the occurrence of side effects) and efficacy (how well the drug works in reducing trigeminal neuralgia attacks) of a drug called lamotrigine in adults with trigeminal neuralgia.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, add-on study of lamotrigine in trigeminal neuralgia. Thirty-eight eligible patients with trigeminal neuralgia will be enrolled; nineteen will be randomized to the active medication group and nineteen to the placebo group. Using a daily diary, all patients will document their overall pain level and attack frequency and intensity for four weeks. After the four week baseline period, patients will initiate medication (lamotrigine or placebo). Patients will titrate until either they reach the maximum dose of 400mg per day and up to 700mg for patients on enzyme-inducing anti-epileptic drugs (EIAED's), their side effects inhibit further increases (known as maximum tolerated dose (MTD)), or their trigeminal neuralgia pain resolves (referred to as pain free dose (PFD)) over eight weeks. Patients will remain on a constant dose of prior medications throughout the study. Patients will remain on maximum dose, MTD, or PFD for a maintenance period of at least eight weeks, and at the end of the maintenance period patients who opt to stay on the medication will be unblinded as to medication and dosage. Primary outcome will be average intensity of daily pain.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 yrs
* Male; or non-pregnant/non-lactating female
* Use of adequate birth-control measures as determined by investigator for females of child-bearing potential
* Diagnosis of trigeminal neuralgia (TN) using IHS (International Headache Society) criteria (see appendix A)
* Able to cooperate with and understand study instructions
* Signed informed consent prior to entering study
* Patients must be on a stable dose of concomitant medications for treatment of trigeminal neuralgia (TN) for at least 4 weeks (see below)
* If subject is currently receiving a tricyclic antidepressant, anticonvulsant, and/or Class I antiarrhythmic (e.g., amitriptyline, mexiletine, phenytoin, gabapentin or carbamazepine) for treatment of pain or any other condition, subject must be willing and able to maintain stable doses of these agents within 4 weeks prior to randomization and throughout the study (i.e., doses cannot be increased or decreased during this period).
* Subjects who require "rescue" analgesic medication during the study will be allowed to use increased doses of their current (pre-study) opioid and/or non opioid analgesics as clinically indicated (e.g., non-steroidal anti-inflammatory medications, acetaminophen, COX-2 inhibitors, topical analgesics). Subjects will be allowed to use a new analgesic for a limited time for non-neuropathic pain (e.g., headache, sinusitis, strained muscle, minor ache and pain), but will be prohibited from initiating therapy with a new analgesic agent and use it continuously throughout the remainder of the study.
* If subject is not currently receiving a tricyclic antidepressant, anticonvulsant, and/or Class I antiarrhythmic (e.g., amitriptyline, mexiletine, phenytoin, gabapentin or carbamazepine) for treatment of pain or any other condition, subject must be willing and able to abstain from initiation of these agents within 4 weeks prior to randomization and throughout the study.
* Subject must be willing and able to abstain from initiating an alternative therapy (e.g., acupuncture, massage or physical therapy) for pain relief during the study. (NOTE: subjects who are currently using alternative therapy for pain relief can be enrolled if they are willing and able to maintain such therapy stable throughout the study.)

Exclusion Criteria:

* Serious hepatic, respiratory, hematologic, cardiovascular or renal condition
* Neurologic pain other than TN (trigeminal neuralgia), with the exception of occasional migrainous/ tension-type headaches. (<4 headaches per month)
* Psychiatric or medical condition that might compromise participation in study, as determined by the investigator
* Use of opioid analgesic as treatment of neuralgia (>2 days per week)
* Administration of any investigational drug within 30 days prior to screening
* Concurrent use of sodium valproate
* Current diagnosis of active epilepsy or any active seizure disorder requiring chronic therapy with antiepileptic drug(s)
* Pregnant or breastfeeding women
* History of substance abuse/ alcoholism

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-06; Primary Completion 2006-05 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlind A Stiles, D.M.D., Principal Investigator — Thomas Jefferson University, Jefferson Headache Center
Locations (1):
- Jefferson Headache Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Lamotrigine: The intervention type is 'drug' and this arm is the active drug supplied by the manufacturers of lamotrigine (Lamictal) to be exact replicas of the actual drug being studied. This drug is an anti-seizure medication.
Period: Overall Study
Arm/Group | Placebo | Lamotrigine
Started | 10 | 10
Completed | 7 | 7
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Lamotrigine: The intervention type is 'drug' and this arm is the active drug created and supplied by the manufacturers of lamotrigine (Lamictal). This is an anti-seizure medication.
- Total: Total of all reporting groups
Arm/Group | Placebo | Lamotrigine | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Pain Attacks
Description: The average number of attacks daily experienced between Visit #1 and Visit #2 (baseline diary) was compared to the average daily number of attacks recorded between Visit #5 and Visit #7 after the patient has titrated the drug to the maximum tolerated dose.
Time Frame: Day 150 Visit #7
Measure: Mean (Standard Deviation); unit: Pain attacks
Arm/Group | Placebo | Lamotrigine
Number analyzed (Participants) | 7 | 7
Pain attacks | 3.3533 (1.1209) | 3.1807 (0.7713)

ADVERSE EVENTS:
Groups:
- Placebo: Subjects who received placebo
- Lamotrigine: Subjects who received Lamotrigine
Arm/Group | Placebo | Lamotrigine
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=7) | Lamotrigine (N=7)
ataxia (Nervous system disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Limited enrollment due to fear of placebo and high drop out rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes